CLINICAL TRIAL: NCT05795387
Title: Add-on Video-based Training: Effect on Mental Status Examination Skills in 5th Year Medical Students - an Educational RCT
Brief Title: Add-on Video-based Training on Mental Status Examination Skills
Acronym: VV-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VV_RCT
Record Dates: First submitted 2023-03-03; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Medical Education
Keywords: e-learning; psychopathology; mental status examination

STUDY DESIGN:
Intervention Model Description: A parallel group, superiority, partial-blinded, cluster-randomized controlled trial where both interventions are an addition to the regular psychiatric clerkship.
Who Masked: Investigator, Outcomes Assessor
Masking Description: As mentioned, it will not be possible to mask students or local lecturers to allocation group. PI receives the clerkship student enrolment list from the faculty, randomize at clerkship location level and merge it with the consent lists collected digitally in SurveyXact. The students that have consented to participation receives individual invitation to the designated e-module. The instructor carrying out the digital mental status examination test, has no information of arm allocation. Statistical analysis will be performed by researcher blind to arm allocation, and masking will only be broken when the primary outcomes have been analyzed and a conclusion has been formulated based on the masked allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Add-on Intervention - Video-based self-regulated training (Experimental): The intervention consist of access to the video e-library on their e-learning platform.
  The video e-library consists of 23 videos of brief patient interviews, mostly with inpatients, with adjoining MSE written by three faculty psychiatrists. Selected videos are used for demonstration of phenomena, and five videos will have audio explanation of the resulting MSE.
  As well as the authentic patient videos on the e-library there are some pages with written theoretical instructions on the MSE, a brief animated movie and some simulated videos by an actor all regarding the MSE.
  Interventions: Other: Video-based self-regulated training on the mental status exam
- Non-video group (Active Comparator): For the present trial, also the NV students will receive the same non-authentic patient material I.E written theoretical instructions on the MSE, a brief animated movie and some simulated videos by an actor all regarding the MSE. Ensuring it is the authentic patient video e-library and not the theoretical information responsible for the expected difference in scores.
  Interventions: Other: E-course with written material on the mental status exam

INTERVENTIONS:
Other: Video-based self-regulated training on the mental status exam — Authentic patient videos for self-regulated training as well as written e-course material, both on the mental status exam
  Arms: Experimental Add-on Intervention - Video-based self-regulated training
Other: E-course with written material on the mental status exam — Written material on the mental status exam
  Arms: Non-video group

SUMMARY:
The goal of this clinical triall is to investigate the training effect of access to authentic patient video on mental status examination performance among 5th year Danish medical students.

Aim:

To investigate if

* Students with add-on access to an authentic patient video e-library have improved Mental Status Examination precision compared to students that only have an add-on e-library with simulated patient videos.
* Number of videos watched correlate to mental status examination test scores.

DETAILED DESCRIPTION:
The main study is a a two-armed, pragmatic cluster-randomised, superiority, partial-blinded, randomized controlled trial where the interventions are e-learning courses that serves as add-on learning material during the psychiatric clerkship.

Two student groups are compared. The experimental intervention(V) is a larger e-learning module, where the students have access to 23 authentic patient video vignettes and an e-module on mental status exam including demonstration videos with simulated patients (actor videos). The comparator students (N-V) only have access to the e-module on mental status exam including demonstration videos with simulated patients. All students participate in the regular Psychiatry curriculum i.e. 16 lectures in one week and psychiatric clerkship in three weeks.

As students have their clerkship in 10 different facilities across the Island of Zealand, we carry out cluster-randomization based on clerkship location.

Communication, recruitment and data management is carried out within the university teaching platform (CANVAS), by manual extraction, and by questionnaires distributed by SurveyXact.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* 5th year medical student at the University of Copenhagen on the psychiatric clinical rotation

Exclusion Criteria:

* Previous acess to the video library.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Mental status exam skills test | A week after the intervention
  The test consists of three subtests each consisting of a video vignette, not accessible in the library (i.e. none of the students had seen it previously) with a forced choice test (FCT). This results in a scoring range of -15 to + 15 points per FCT. The MSE-skills test score consists of the student's average score of the three FCTs.

SECONDARY OUTCOMES:
MSE skill test score stratification | Baseline
  We will explore if there is a difference between gender, each individual video and attitude towards psychiatry on the MSE skill test score
General evaluation of the clinical rotation | Immediately after the intervention
  The evaluation is carried out by a validated questionnaire of 10 items, to be answered on a 5-point Likert scale. Purpose-made supplementary questions concerning the student's number of patient encounters alone and with a doctor/staff and area of interest in psychiatry
Questions concerning use of the video e-library | Immediately after the intervention
  time spend on each task/video ; evaluation of/satisfaction with the different element of the e-library

CONTACTS AND LOCATIONS:
Overall Officials: Sidse M Arnfred, Professor, Study Director — Research Unit Psychotherapy and Psychopathology Psychiatry West; Esben B Schäfer, MD, Principal Investigator — Research Unit Psychotherapy and Psychopathology Psychiatry West
Locations (2):
- Denmark (2):
  - Mental Health Service Capital Region, Copenhagen
  - Mental Health Service Region Zealand, Slagelse

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT05795387/Prot_000.pdf